CLINICAL TRIAL: NCT03440151
Title: Oncological Outcome of Contralateral Submental Artery Island Flap Versus Primary Closure in Tongue Squamous Cell Carcinoma (Randomize Noninferiority Clinical Trial)
Brief Title: Oncological Outcome of Contralateral Submental Artery Island Flap Versus Primary Closure in Tongue Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omer mohammed jamali, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 513
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Tongue Squamous Cell Carcinoma
Keywords: Tongue Squamous Cell Carcinoma,; Contralateral Submental Flap; Submental Flap; oncological safety

STUDY DESIGN:
Masking Description: Because the two interventions used in this trial are clearly different and easly recognized by the participants and investigators, neither investigators nor Participants can be blinded.
  The statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contralateral submental flap for tongue cancer defect (Experimental)
  Interventions: Procedure: contralateral submental flap for tongue cancer defect
- primary closure for tongue cancer defect (Active Comparator)
  Interventions: Procedure: primary closure for tongue cancer defect

INTERVENTIONS:
Procedure: contralateral submental flap for tongue cancer defect — Tumor resection will be star first this accomplish with 1- 2 cm safety margin, Simultaneous neck dissection will be performed in all patient.
  Flap dissection begins from the opposite side of the pedicle in the subplatysmal plane. Then the level 1a is dissected, the distal facial artery and facial vein to the branching point of the submental pedicle are ligated. The anterior belly of the digastric muscle on ipsilateral to the pedicle and strip of mylohyoid muscle will dissected off the mandible and the hyoid bone and included with the flap. This results in complete mobilization of the flap.A tunnel will be created between the defect and the donor site and the skin paddle of the flap will be transported through it intraorally and the flap is insetted.
  Arms: contralateral submental flap for tongue cancer defect
Procedure: primary closure for tongue cancer defect — Under general anesthesia the tumor will be resected with Preserving floor of mouth mucosa as much as possible to avoid restriction of tongue mobility. After Obtaining meticulous hemostasis, the tongue defect will be closed in layers.
  Arms: primary closure for tongue cancer defect

SUMMARY:
The purpose of this study is to compare the oncological and functional results of the contralateral submental flap with primary closure for reconstruction of tongue squamous cell carcinoma.

DETAILED DESCRIPTION:
Resection of tongue malignancies remains one of most surgical challenges because of its adverse effects on speech articulation, swallowing, and eventual quality of life.

A variety of local flaps such as infrahyoid flap and the Platysma flap, and free flaps like the radial forearm and anterolateral thigh (ALT) flap have been available for reconstruction of tongue. However, all these options have their shortcomings.

When reconstructing particular oral cavity defect the tissue used should be reliable; functional and cosmetically acceptable with minimum donor site morbidity and match the recipient site in terms of color, texture and thickness. The submental island flap (SMI-flap) which has been first introduced by Martin et al in 1990, meets all these requirements and due to its optimal location, ease of harvest, and favorable arc of rotation, the SMI-flap has gained acceptance as a simple, reliable and convenient to repair defects of tongue and oral cavity cancer.

The oncological safety of submental flap in oral cancer patient still debate, this is due to its proximity to the main nodal basins of levels 1A and 1B and the possibility of transfer of occult metastatic lymph node to the recipient site during reconstruction.

in addition some authors has not been recommended submental flap for cases with clinically or radiologically established nodal disease as it might compromise the oncological resection and continuity of neck dissection and so alternative options should be considered. The contralateral submental island flap (CSMI-flap) is believed to offer such alternate option for patient with contralateral negative node.

our a priori-hypothesis is that utilization of the CSMI-flap is not related to an altered prognosis in tongue squamous cell carcinoma patients. In order to test this hypothesis, we will compare the oncological outcome of group of patients receive CSMI-flap with the results of another group of patients not receive CSMI-flap and close tongue defect by primary closure, which is another well-established concept of management tongue cancer defect.

ELIGIBILITY:
Inclusion Criteria:

* Patient with T1&T2 tongue squamous cell carcinoma.

Exclusion Criteria:

* Patients with contralateral N positive.
* Patients with previous neck surgery that interrupt contralateral facial artery or vein.
* Patients with prior radiotherapy to the neck.
* Patients with lesions crossing the midline, or those reaching the base of tongue requiring total glossectomy.
* Patients second primary tumors at the time of diagnosis.
* Patient with recurrent tongue squamous cell carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
local recurrence | at least one year post operative

CONTACTS AND LOCATIONS:
Overall Officials: Omer M Jamali, phd student, Principal Investigator — Cairo University
Locations (1):
- Omer M Jamali, Cairo, Faculty of Dentistry-Cairo University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided